CLINICAL TRIAL: NCT03683706
Title: Feasibility Trial of Learning Through Play (LTP) in My Own Way Plus CBT A Parent-Based Intervention for Depressed Mothers With ID Children
Brief Title: Learning Through Play (LTP) in My Own Way Plus CBT
Acronym: Umeed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: LTP In My Own Way Plus
Record Dates: First submitted 2018-09-19; First posted 2018-09-25 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Intellectual Disability; Depression
MeSH Terms: conditions — Intellectual Disability; Depression | interventions — Long-Term Potentiation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Researchers doing outcome assessments will be kept blind to treatment allocations
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Participants in this arm will receive 12 sessions of LTP in My Own Way Plus interventions.
  Interventions: Behavioral: LTP in My Own Way Plus
- Treatment as Usual (No Intervention): Participants in this arm will be getting their usual treatment

INTERVENTIONS:
Behavioral: LTP in My Own Way Plus — LTP in My Own Way Plus is a 12-session integrated intervention-Learning through Play in My Own Way Plus Cognitive Behaviour Therapy (CBT). LTP in My Own Way is the extension of the parent education program called 'Learning Through Play' developed by Toronto Public Health (1993) revised by The Hincks-Dellcrest Centre (2000). LTP aims for the healthy growth of young children (birth to 6 years) using the stages of development incorporating Piaget's theory of cognitive development and Bowlby's theory of attachment. The objective of this program is to strengthen parent-child attachment by encouraging parental involvement and teaching parents how to use play activities to enhance their children's development. Second component of intervention is CBT adapted from Jeanne Miranda manual (Group CBT for Depression, group leaders guide book-2006) focusing on the three areas: thoughts and your mood, activities and your mood, people interaction and your mood.
  Arms: Intervention

SUMMARY:
Aim of the study is to evaluate the acceptability and feasibility of LTP in My Own Way Plus with depressed mothers of ID children.

DETAILED DESCRIPTION:
Having a child with a chronic medical problem or an intellectual disability increases anxiety and depression in parents. There is some growing evidence that families of ID children are able to meet the challenges. The purpose of the present study is to adapt LTP in my own way plus to test its acceptability and determine if it improves mothers knowledge about their child development and reduce their level of distress.

The study has two phases: quantitative phase and qualitative phase. Quantitative phase: A single blind randomised controlled trial in school settings in Karachi Pakistan.

Objectives:

1. Help mothers cope better with their depression.
2. Teach mothers play activities that will stimulate their children's development and improve mother-child interaction.

Qualitative Phase: This will help to determine acceptability of the intervention and identify perceived mechanisms of change and any barriers and facilitators to LTP in my own Plus intervention. In-depth digitally recorded interviews and focus groups will be conducted with the parents and teachers to understand their beliefs, views, and feelings about caring for ID children.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of ID children aged 3 to 6 years, screened positive for depression
* Ability to complete a baseline assessment
* Ability to communicate in Urdu or English

Exclusion Criteria:

* Have a diagnosed serious medical or psychiatric condition
* Mothers of children with other medical illness
* Temporary residents unlikely to be available for follow-up

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2020-10-08 (Actual)

PRIMARY OUTCOMES:
Session Log (Feasibility and acceptability) | change in baseline to 12 weeks
  sessions logs (attendance of each participant) will be maintained.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) (Kroenke, Spitzer, & Williams, 2003): | change in baseline to 12 weeks
  The Patient health Questionnaire (PHQ-9) is 10 items self-report questionnaire for screening, diagnosing and measuring severity of depression which is easy to use and can be administered by a trained research worker. Score ranges from 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.
Generalized Anxiety Disorder (GAD) 7 (Spitzer, Kroenke, Williams, & Löwe, 2006): | change in baseline to 12 weeks
  The GAD-7 is a 7-item scale used to screen for and measure severity of generalized anxiety disorder. Scores of 5, 10 & 15 are taken as cut-off points for mild, moderate and high. it takes about 5 minutes to administer this sca
Vineland Adpative Behaviour Scales (VABS-II) VABS-II (Sparrow et al., 2005): | change in baseline to 12 weeks
  VABS-II measure adaptive behaviors of individuals from birth to 90 years. The main domains are communication, daily living skills, socialization, and motor skills. The parent/caregiver self-report form requires a completion time of 30-60 minutes and yields an adaptive behaviour composite score.

CONTACTS AND LOCATIONS:
Overall Officials: Nasim Chaudhry, Principal Investigator — Pakistan Institute of Living & Learning
Locations (1):
- A private school in Karachi, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No